CLINICAL TRIAL: NCT06218680
Title: Efficacy of Low Dose Propofol Given at the End of Sevoflurane Anesthesia for Prevention of Emergence Agitation in Pediatric Patient Undergoing MRI Scan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Santhita Pimonbut, Santhita Pimonbut, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HE661348
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Saline Solution

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group P (Experimental): Receive 0.5 mg/kg of propofol intravenously at end of sevoflurane anesthesia
  Interventions: Drug: Propofol
- group S (Placebo Comparator): Receive saline intravenously at end of sevoflurane anesthesia
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Propofol — recieve propofol 0.5 mg/kg intravenously at end of sevoflurane anesthesia
  Arms: group P
Drug: Normal saline — recieve propofol 0.5 mg/kg intravenously at end of sevoflurane anesthesia
  Arms: group S

SUMMARY:
The goal of this clinical trial is to compare Efficacy of low dose propofol(0.5 mg/kg) vs placebo given at the end of sevoflurane anesthesia for prevention of emergence agitation in pediatric patient undergoing MRI scan. The main question it aims to answer is "Can low dose propofol reduce the incidence of emergence agitation after general anesthesia?" Participants will be given propofol 0.5 mg/kg or saline according to the allocated group at the completion of MRI scan

ELIGIBILITY:
Inclusion Criteria:

* Age 2-8 years
* ASA class I or II ,who schedule for MRI scan under sevoflurane anesthesia

Exclusion Criteria:

* Developmental delay
* Psychological and neurological disorders
* Abnormal airway
* Reactive airway disease
* Allergy to propofol, egg product
* Family history of malignant hyperthermia
* Need iv sedative medication before induction
* Obesity

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
incidence of emergence agitation | at 5,10,15,20,25,30 minutes after extubation

SECONDARY OUTCOMES:
Incidence of complication | 2 hours after extubation
  Nausea or vomiting, airway obstruction, laryngospasm, desaturation and apnea
Use of rescue medication | 2 hours after extubation
  use of ondansetron, atropine
Emergence time | 2 hours after extubation
  duration of emergence
Length of stay in post anesthetic care unit | 2 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Santhita Pimonbut, M.D., Principal Investigator — department of anesthesiology, faculty of medicine, Khonkaen University
Locations (1):
- Khon kaen University, Khon Kaen, Muang, Thailand

IPD SHARING:
Plan to Share IPD: Yes
all collected individual participant data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 month after publication
Access Criteria: Researcher who required more information for further study

REFERENCES:
- [Background] Kulka PJ, Bressem M, Tryba M. Clonidine prevents sevoflurane-induced agitation in children. Anesth Analg. 2001 Aug;93(2):335-8, 2nd contents page. PMID 11473855
- [Background] Welborn LG, Hannallah RS, Norden JM, Ruttimann UE, Callan CM. Comparison of emergence and recovery characteristics of sevoflurane, desflurane, and halothane in pediatric ambulatory patients. Anesth Analg. 1996 Nov;83(5):917-20. doi: 10.1097/00000539-199611000-00005. PMID 8895263
- [Background] Aouad MT, Yazbeck-Karam VG, Nasr VG, El-Khatib MF, Kanazi GE, Bleik JH. A single dose of propofol at the end of surgery for the prevention of emergence agitation in children undergoing strabismus surgery during sevoflurane anesthesia. Anesthesiology. 2007 Nov;107(5):733-8. doi: 10.1097/01.anes.0000287009.46896.a7. PMID 18073548
- [Background] Cravero JP, Beach M, Thyr B, Whalen K. The effect of small dose fentanyl on the emergence characteristics of pediatric patients after sevoflurane anesthesia without surgery. Anesth Analg. 2003 Aug;97(2):364-367. doi: 10.1213/01.ANE.0000070227.78670.43. PMID 12873918
- [Background] Costi D, Ellwood J, Wallace A, Ahmed S, Waring L, Cyna A. Transition to propofol after sevoflurane anesthesia to prevent emergence agitation: a randomized controlled trial. Paediatr Anaesth. 2015 May;25(5):517-23. doi: 10.1111/pan.12617. Epub 2015 Jan 13. PMID 25586124
- [Background] Ramlan AAW, Pardede DKB, Marsaban AHMS, Hidayat J, Peddyandhari FS. Efficacy of 0.5 mg/kg of propofol at the end of anesthesia to reduce the incidence of emergence agitation in children undergoing general anesthesia with sevoflurane. J Anaesthesiol Clin Pharmacol. 2020 Apr-Jun;36(2):177-181. doi: 10.4103/joacp.JOACP_257_19. Epub 2020 Jun 15. PMID 33013031
- [Background] Abu-Shahwan I. Effect of propofol on emergence behavior in children after sevoflurane general anesthesia. Paediatr Anaesth. 2008 Jan;18(1):55-9. doi: 10.1111/j.1460-9592.2007.02376.x. PMID 18095967